CLINICAL TRIAL: NCT02403583
Title: Jamii Bora: A Home-based Couples Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Kenya Medical Research Institute (Other); University of California, San Francisco (Other); National Institute of Mental Health (NIMH) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Janet M. Turan, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: X140304009; 1R34MH102103-01A1 (NIH)
Record Dates: First submitted 2015-02-24; First posted 2015-03-31 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV Transmission; Prevention of Mother to Child Transmission; Serodiscordancy; Home-based testing; Home-based counseling; Linkage to care; Couples HIV Testing and Counseling; Acceptance of repeat HIV testing during pregnancy; Retention in care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention- Home visits (Other): Participants randomized to intervention arm receive 3 home visits conducted by one female and one male lay health worker.
  Interventions: Behavioral: Intervention- Home Visits
- Standard Care (No Intervention): Participants will receive current standard clinic-based services including the option for women and partners to return to the clinic for male partner HIV testing or CHCT.

INTERVENTIONS:
Behavioral: Intervention- Home Visits — If a woman has been randomized to the intervention arm, a lay health worker will obtain detailed locator information (including cell phone contacts) and consult with the woman about optimal times for a home visit. The woman will be given a letter for her male partner to inform him about the study and potential upcoming visits, given that our preliminary research revealed that notifying the male partner beforehand is important. As described above, the intervention arm will consist of three home visits conducted by one female and one male lay health worker.
  Arms: Intervention- Home visits

SUMMARY:
The purpose of the study is to develop and pilot-test a home-based intervention to facilitate sate HIV testing and disclosure within pregnant couples in order to increase use of prevention-of-mother-to-child-transmission (PMTCT) and family health services in Kenya.

DETAILED DESCRIPTION:
Despite the potential for anti-retroviral therapy (ART) to ensure maternal health and reduce vertical HIV transmission to as low as 1%, HIV-related maternal deaths and HIV infection among infants remain unacceptably high across sub-Saharan Africa. Prevention of mother-to-child transmission (PMTCT) requires a complex series of interventions throughout pregnancy and after birth, and only an estimated 15-30% of eligible women complete this "PMTCT cascade". Drop-offs can occur in the PMTCT cascade if women refuse HIV testing, do not disclose their HIV status, or avoid essential health services because they fear negative consequences for their relationship with their male partner. Engaging both partners of a couple during pregnancy has the potential to enhance health decisions, increase healthcare utilization, and ultimately improve maternal, paternal, and infant health. The goal of this study is to develop and pilot a home-based couples intervention that includes safe HIV testing and disclosure for couples, alongside information and counseling for family health during the perinatal period. The investigators will adapt existing evidence-based Couples HIV Counseling and Testing (CHCT) protocols for the special needs of pregnant women and their male partners, and train pairs of lay health workers (one female and one male) to deliver this service as part of home visits in rural Kenya. As men rarely attend antenatal clinics in Kenya, a home-based strategy can reach the couple in a safe and convenient space and give them unprecedented access to family health information, CHCT services, and linkage to care. This intervention, based on an interdependence model of communal coping and behavior change, is expected to help couples to communicate, plan, and take action around HIV and family health. Building on our team's preliminary studies in this rural Kenyan setting, the investigators collected further formative data and translated our findings into a viable intervention model with input from local stakeholders. The investigators will then conduct a pilot study of the home-based couples intervention, in which the investigators will randomize pregnant women at two antenatal clinics to the intervention or standard care arms of the study, and follow them and their male partners until three months after the expected delivery date of the baby. The investigators will preliminarily assess the effects of the intervention on uptake of CHCT by couples, repeat HIV testing during pregnancy for HIV-negative women, and utilization of PMTCT and HIV services for HIV-positive women and men. The investigators will also explore the roles of potential mediators for these effects suggested by our interdependence conceptual framework (such as measures of couple relationship dynamics). Results from this study will provide evidence of the preliminary impact, acceptability, and feasibility of the intervention and the study methods that will allow our team to develop a larger-scale efficacy trial. Engaging pregnant couples in family health and PMTCT is an essential step towards reducing HIV-related maternal mortality and eliminating new HIV infections among children in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* (a) 18 years of age or older (b) 36 weeks of pregnancy or less (c) has been offered HIV testing at ANC, (d) is currently in a stable relationship (married or cohabiting) with a male partner of duration of at least 6 months (e) is currently living with a male partner who will be in residence at least one night a week at the home during the study period, (f) has not yet participated in couple HIV counseling and testing during this pregnancy (g) has not disclosed current HIV status to male partner (h) does not know with certainty the HIV-positive status of her male partner.

Exclusion Criteria:

* (a) Currently pregnant (b) Greater than 36 weeks of pregnancy (c) Less than 18 years of age (d) Not currently in a stable relationship of at least 6 months (e) Does not currently live with male partner at least one night a week at the home (f) Has not been offered HIV testing (g) Has received CHCT with current male partner (h) has disclosed current HIV status to male partner (i) Knows with certainty current male partner is HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Utilization of maternal and child health (MCH) services (outcome for all couples in the study) | 3 months after the expected due date of the baby
  Composite variable including at having completed least four antenatal care (ANC) visits during pregnancy (Y/N), childbirth with a skilled attendant (Y/N), and postnatal check-ups for woman (Y/N) and infant (Y/N). These are assessed in the follow-up questionnaire completed at three months after the baby's estimated due date.
Use of PMTCT interventions (for HIV+ women only) | 3 months after the expected due date of the baby
  Composite variable including mothers use of antiretrovirals (ARVs) (Y/N), prophylactic ARVs given to the infant (Y/N), and appropriate infant feeding mode (Y/N). These are assessed in the questionnaire completed at three months after the baby's estimated due date.

OTHER OUTCOMES:
Couple HIV testing (all couples) | 3 months after the expected due date of the baby
  CHCT Uptake (Y/N) - This variable is coded Yes if the couple accepts and undertakes CHCT during the observation period (up to three months after the expected due date of the baby). This is assessed at each couple visit.
Antenatal HIV testing (outcome for women who initially tested HIV-negative) | 3 months after the expected due date of the baby
  Re-testing for HIV during pregnancy. This is assessed in the questionnaire completed three months after the baby's estimated due date.

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Turan, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- Kenya (5):
  - Macalder District Hospital, Migori, Migori County
  - Oyani Health Center, Migori, Migori County
  - Wath Onger, Othoch Rakuom, Migori County
  - Rongo District Hospital, Rongo, Migori County
  - God Jope Dispensary, Suna, Mirgori

REFERENCES:
- [Derived] Turan JM, Darbes LA, Musoke PL, Kwena Z, Rogers AJ, Hatcher AM, Anderson JL, Owino G, Helova A, Weke E, Oyaro P, Bukusi EA. Development and Piloting of a Home-Based Couples Intervention During Pregnancy and Postpartum in Southwestern Kenya. AIDS Patient Care STDS. 2018 Mar;32(3):92-103. doi: 10.1089/apc.2017.0285. PMID 29620927